CLINICAL TRIAL: NCT04193787
Title: Expanding PrEP Implementation in Communities of People Who Inject Drugs and Their Risk Network Members
Brief Title: EPIC-P Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Roman Shrestha, Assistant Professor, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E20-0594
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EPIC-P (Experimental): Participants will enroll in a bio-behavioral intervention aimed at preventing HIV transmission in people who inject drugs.
  Interventions: Other: EPIC-P

INTERVENTIONS:
Other: EPIC-P — EPIC-P is a brief, bio-behavioral intervention based on the information-motivation-behavioral skills (IMB) model framework, which integrates i) a biomedical component (i.e., PrEP), ii) behavioral components (i.e., drug- and sex-related primary HIV prevention), and iii) mHealth technology (i.e., text messaging PrEP reminders).

SUMMARY:
This non-randomized, open-label study will address the following research aims in People who inject drugs (PWID):

* To assess the feasibility and acceptability of the Expanding PrEP Implementation in Communities of PWID (EPIC-P) intervention among high-risk PWID.
* To determine the preliminary efficacy of the EPIC-P intervention in terms of increasing adherence to PrEP and primary HIV prevention among high-risk PWID.

DETAILED DESCRIPTION:
A non-randomized, open-label design will be utilized to test the feasibility, acceptability, and preliminary efficacy of the Expanding PrEP Implementation in Communities of PWID (EPIC-P) intervention among high-risk people who inject drugs (PWID) with opioid dependence (N=100). Since the aim of this pilot study is to establish whether the EPIC-P intervention is feasible/acceptable among at-risk PWID in a community-based setting, proposed is a non-comparative design. With the hopes to target PWID who are not linked with existing harm reduction services, proposed is to recruit participants using respondent driven sampling (RDS), a chain referral method with demonstrated success in recruiting hard-to-reach populations. Initial RDS participants, called "seeds," will be carefully recruited from the community where the study team leadership have built a well-established relationship. Participants enrolled in the study will be assessed at baseline and will be followed for 9 months (with follow-up assessments at 3- and 6-months) by trained research assistants. Importantly, structured interviews will be conducted at follow-up visits to examine the barriers and facilitators and feedback about optimal implementation of the EPIC-P intervention.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the Greater New Haven area;
* Confirmed HIV-negative;
* Reporting injection drug use (past 3 months) with substantial ongoing risk for HIV acquisition;
* Started on PrEP (within the last week).

Exclusion Criteria:

* Not on PrEP;
* Not available during the full duration of the study;
* Cannot speak English;
* Unable to provide consent;
* Anyone actively suicidal, homicidal, or psychotic as assessed by trained research staff under the supervision of a consultant that is a licensed clinical psychologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Retention Rate | Up to 6 months
  To determine feasibility, the rate of enrolled participants that are retained through the study will be assessed.

SECONDARY OUTCOMES:
Acceptability | Up to 6 months
  The acceptability will be assessed using a series of eight items acceptability rating profile. We will use a 5-point Likert scale (0= strongly disagree to 4= strongly agree) to rate the extend to which they agreed with each acceptability statement. A mean intervention acceptability score will be calculated with higher values indicating greater acceptability.
PrEP Adherence VAS | Up to 6 months
  Adherence to PrEP will be assessed using a visual analog scale (VAS).
PrEP Adherence Pharmacy | Up to 6 months
  Adherence to PrEP will be assessed by monitoring the pharmacy refills of participants.
PrEP Adherence DBS | Up to 6 months
  PrEP Adherence will be objectively assessed using dried blood spot (DBS) testing for tenofovir levels.
HIV Incidence | Up to 6 months
  HIV incidence will be tracked in participants through testing up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Shrestha, PhD, MPH, Principal Investigator — Associate Research Scientist, Yale School of Medicine
Locations (1):
- Storefront, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gautam K, Paudel K, Wickersham JA, Altice FL, Bellia G, Jadkarim L, Liew Z, Khati A, Copenhaver M, Shrestha R. Feasibility and acceptability of daily oral emtricitabine/tenofovir alafenamide fumarate (FTC/TAF) for HIV pre-exposure prophylaxis among people who inject drugs with opioid use disorder. Sex Transm Infect. 2026 Feb 10:sextrans-2025-056770. doi: 10.1136/sextrans-2025-056770. Online ahead of print. PMID 41667236